CLINICAL TRIAL: NCT05308784
Title: A Survey of Physician and Molecular Tumor Board Perspectives on the Clinical Utility and Usability of Cellworks Singula™ and Ventura™ Reports in Facilitating Patient Treatment Decisions for Pan-Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Avera McKennan Hospital & University Health Center (Other)
Collaborators: Cellworks Group Inc. (Industry)
Responsible Party: Principal Investigator, Tobias Meissner, Manager -- Cancer Genomics, Avera McKennan Hospital & University Health Center
Other Study IDs: myCare-101
Record Dates: First submitted 2022-03-21; First posted 2022-04-04 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Pan-cancer

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Cellworks Singula and Ventura reports — Personalized drug match reports based on patients' genomic aberration.

SUMMARY:
The purpose of this study is to determine the benefit of Cellworks Singula™ and Ventura™ reports on physician and molecular tumor board treatment recommendations across a large set of pan-cancer indications. Cellworks reports aim to provide NGS-based therapy recommendations to aid the decision-making of patients, physicians, and molecular tumor boards.

ELIGIBILITY:
1. Have any stage of cancer for the indications listed at: https://cellworks.life/mycare101 Patients are eligible at any stage of disease.
2. Expected to be alive 6 months or more
3. Requirements for NGS testing (e.g., panel or whole-exome sequencing): NGS testing has been ordered from or performed by one or more vendors specified at: https://cellworks.life/mycare101 . NGS reports must be ordered or performed within the last 90 days. Cellworks will accept all NGS input formats available, including PDF, VCF, BAM, and FastQ.
4. Requirements for additional laboratory testing If Hematological Indication, Cytogenetics in the form of FISH, Karyotyping, IHC, and/or aCGH has been ordered If Acute Myeloid Leukemia (AML), FLT3-itd testing has been ordered If Indication is a form of Brain Cancer (e.g., glioblastoma), Cytogenetics in the form of FISH, Karyotyping, IHC, and/or aCGH has been ordered and MGMT Methylation test has been ordered

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a diagnosis of cancer at any stage
Sampling Method: Probability Sample
Enrollment: 730 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Physician satisfaction on Cellworks reports | 2022.1 - 2023.1
  A questionnaire will be administered following receipt of the Cellworks report. Survey questions will be performed using a 6-point forced response Likert scale. Simple descriptive statistics, including medians, mode and range of the resulting Likert scores, will be reported but can lead to incorrect effect size estimates, inflated error rates, and other issues (Bürkner & Vuorre, 2019).
  For hypothesis testing purposes, the proportion of physicians and MTB's with a favorable response (i.e., Likert score of 4 or above) will be estimated along with exact (Clopper-Pearson) 95% two-sided confidence intervals.

CONTACTS AND LOCATIONS:
Locations (1):
- Avera McKennan, Sioux Falls, South Dakota, United States